CLINICAL TRIAL: NCT06544629
Title: Imjudo & Imfinzi Post-Marketing Surveillance
Brief Title: Imjudo & Imfinzi PMS
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D419CR00029
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Based on the re-review of new drugs article, Korean pharmaceutical act, the objectives of this study are to assess safety and effectiveness of the study drugs(Imjudo & Imfinzi) in a real world setting in patients who treated according to the approved indications in Korea.

DETAILED DESCRIPTION:
Primary Objective:

To assess safety of the study drugs for patients treated with the study drugs under the approved indication in Korea

Secondary Objective:

To assess effectiveness of the study drugs for patients treated with the study drugs under the approved indication in Korea

Exploratory Objective:

To assess effectiveness of the study drugs for patients treated with the study drugs under the approved indication in Korea

ELIGIBILITY:
Inclusion criteria:

1. Patients eligible for the study drugs according to the approved label in Korea
2. Provision of signed and dated written informed consent by the patient or legally acceptable representative

Exclusion criteria:

1. Other off-label indications according to the approved label in South Korea
2. Current participation in any interventional trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who initiate treatment with study drugs after the contract date for the first time.
Sampling Method: Non-Probability Sample
Enrollment: 246 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Safety (adverse events (AEs), serious AEs (SAEs), adverse drug reactions (ADRs), serious ADRs (SADRs), unexpected AEs/ADRs) | For Imjudo will be conducted for 90 days from the first dose of the treatment. For Imfinzi will be separately conducted for 1 year from the first dose.
  To assess safety of the study drugs for patients treated with the study drugs under the approved indication in Korea

SECONDARY OUTCOMES:
Objective Response Rate(ORR) | For 1 year from the first dose of the treatment
  To assess effectiveness of the study drugs for patients treated with the study drugs under the approved indication in Korea

OTHER OUTCOMES:
Disease Control Rate (DCR) | For 1 year from the first dose of the treatment
  To assess effectiveness of the study drugs for patients treated with the study drugs under the approved indication in Korea

CONTACTS AND LOCATIONS:
Locations (5):
- South Korea (5):
  - Research Site, Busan
  - Research Site, Goyang
  - Research Site, Seongnam
  - Research Site, Seoul
  - Research Site, Suwon